## Alabama Healthy Marriage and Relationship Education Initiative Informed Consent Letter

February 27, 2020 NCT03158714



## NOTE: DO NOT SIGN THIS DOCUMENT UNLESS AN IRB APPROVAL STAMP WITH CURRENT DATES HAS BEEN APPLIED TO THIS DOCUMENT.

## INFORMATION AND CONSENT LETTER

For the "Alabama Community Healthy Marriage Initiative" Couples Evaluation Project **Participant** 

You are invited to participate in an evaluation project focused on the effectiveness of marriage and relationship education programs. This project is being conducted by Dr. Francesca Adler-Baeder from the Department of Human Development and Family Studies and Dr. Christine Totura from the Department of Psychology at Auburn University. We hope to learn about the effectiveness of Healthy Marriage and Relationship Education (HMRE) programs on building individual, couple, and family strengths. We also hope to learn about general impressions of the programs, the facilitators, and suggestions for ways to improve the program. This information will help us verify if the programs are meeting their objectives and will help us make improvements to the design of the programs that can improve their effectiveness for families like yours in this community and others around the state and nation. This information may also be used to develop presentations and journal articles for professional meetings and publications. You are invited to participate because of your interest in receiving programming and because you are age 19 or older and are in a committed couple relationship.

What will be involved if you participate? All couples interested in programming will be eligible to participate in this local impact evaluation, a randomized control trial (RCT) that will be used to evaluate HMRE classes on marriage and couple functioning. As a couple, you will be randomly assigned (much like the flip of a coin) using a unique couple ID to either participate in a 6-week HMRE class (ELEVATE or Couples Connecting Mindfully) or to be part of the comparison group which does not participate in a class during the evaluation project period. For all groups, couples will be asked to individually complete a series of online surveys: one before the programs start, one immediately after completion of the program, one at 6 months and one at 1-year and 2-year followups. Each survey is expected to take an average of 60 minutes to complete, and the surveys will assess individual, couple, and family relationship characteristics, as well as attitudes and beliefs about programming if you are assigned to a class.

Are there any risks or discomforts? Some of the questions may be sensitive in nature, and it may be somewhat uncomfortable to answer them. You do not have to answer any question that you do not want to. You may withdraw from participation at any time, without penalty, and vou may withdraw any identifiable data that has been collected about you. Your decision whether or not to participate will not affect your current or future relations with Auburn University or the agency delivering the programs.

Are there any benefits? All couple participants in the evaluation project will be compensated in tiered levels. Participants will receive \$50 for completing each of the following surveys: preprogram, immediate post-test if you participate in a program or 6-8 weeks after the first survey if you are in the comparison group, 6-month follow-up, 1-year follow-up. At the 2- year follow-up, participants will receive \$100 for completing the surveys. In total, you are eligible to individually receive \$300 over the 2 years if you complete all 5 surveys.

| Participant's Initials |
|------------------------|
|------------------------|

**The Auburn University Institutional Review Board has approved this Document for use from** 08/07/2017 to 08/14/2018 16-248 EP 1608 Protocol #

Your privacy will be protected. All of the information that you provide on the surveys will be treated as private and kept confidential. Your name will not appear on any surveys. You will be assigned a code number, which will be used to organize the information you provide. Dr. Adler-Baeder and eligible research staff will maintain the enrollment database that shows which number is assigned to you. This information will be kept separate from your completed surveys. To help us further protect your privacy, we have obtained a legal document called a Certificate of Confidentiality from the National Institute of Health. Dr. Adler-Baeder can use this Certificate to legally refuse to disclose information that may identify you, even by a court subpoena in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. Dr. Adler-Baeder will use the Certificate to resist any demand for information that would identify you. If you give someone or an organization written permission to see the information you gave Dr. Adler-Baeder, we cannot use the Certificate of Confidentiality to protect your information from that person or organization.

When would your information have to be shared? If we learn that you or someone else is harming you, your child, or others around you, we may be required to report this to the police or a social service agency in your community, as we are legally required to report violations of Alabama's Child Abuse and Neglect laws. If results of the evaluation are published in a journal, no names of individuals will be included in these reports. All data and results are reported for the group of participants in the evaluation project.

If you have any questions we invite you to contact our research team at (334)-844-8711. If you have questions later, Dr. Adler-Baeder (at (334)-844-4151 or <u>adlerfr@auburn.edu</u>) or Dr. Christine Totura (at (334)-844-4412 or cwt0006@auburn.edu) will be happy to answer them. You will be provided a copy of this form to keep.

For more information regarding your rights as a research participant you may contact the Auburn University Office of Human Subjects Research or the Institutional Review Board by phone (334)-844-5966 or e-mail at <a href="https://hsubjec@auburn.edu">hsubjec@auburn.edu</a> or <a href="https://hsubjec@auburn.edu">IRBChair@auburn.edu</a>.

HAVING READ THE INFORMATION PROVIDED, YOU MUST DECIDE IF YOU WANT TO PARTICPATE IN THIS RESEARCH AND THE RANDOMIZED CONTROL TRIAL EVALUATION PROJECT. IF YOU DECIDE TO PARTICIPATE, THE DATA YOU PROVIDE WILL SERVE AS YOUR AGREEMENT TO DO SO.

| Participant's signature | Date | Investigator's signature I |
|---|---|---|
| | | Dr. Francesca Adler-Baeder |
| Printed name of participant | | Printed name of Investigator |
| The Auburn University Institutional Review Board has approved this Document for use from 08/07/2017 to 08/14/2018 | | Co-Investigator's signature |
| Protocol # 16-248 EP 1608 | | Dr. Christine Totura |
| | _ | Printed name of Co-Investigator |

\_\_\_\_\_ to \_\_\_\_\_. Protocol #\_\_\_\_\_